CLINICAL TRIAL: NCT01351389
Title: Brief Interventions in the Emergency Department for Alcohol and HIV/Sexual Risk
Acronym: SAFER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Memorial Hospital of Rhode Island (Other); Kent Hospital, Rhode Island (Other)
Responsible Party: Principal Investigator, Peter Monti, Professor, Brown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2R01AA009892-16A1 (NIH); 2R01AA009892-16A1 (NIH)
Record Dates: First submitted 2011-05-09; First posted 2011-05-10 (Estimated); Results first posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Alcohol Consumption; Unsafe Sex
Keywords: Brief; Alcohol; Intervention; Sex; Risk
MeSH Terms: conditions — Alcohol Drinking; Unsafe Sex; Coitus | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brief Motivational Intervention (BMI) (Active Comparator)
  Interventions: Behavioral: Brief Motivational Intervention (BMI)
- Brief Advice (Active Comparator)
  Interventions: Behavioral: Brief Advice

INTERVENTIONS:
Behavioral: Brief Motivational Intervention (BMI) — The BMI incorporates open-ended exploration, personalized feedback, and discussion about patients' alcohol use and sexual behaviors and the consequences of these behaviors. Using the central principles described by Miller and Rollnick (2002), the goal of the session, conducted in the hospital as soon as possible, is to explore the patient's alcohol use and sexual behaviors and to help patients consider what they might want to change. Also included is a presentation of personalized feedback, and for patients who are interested in change, a focus on establishing goals for reduced drinking and sexual risk abstinence. Collaboratively the counselor and patient develop a plan for the future, identify goals for behavior change, explore barriers to changes, and provide strategic advice.
  Other Names: BMI
  Arms: Brief Motivational Intervention (BMI)
Behavioral: Brief Advice — Patients in the Brief Advice (BA) condition will receive intervention consistent with standard medical practice when alcohol problems or sex-risk behaviors are indicated. Project staff will offer BA about level of alcohol/drug and sexual behaviors and drug problems risk, and will provide a list of treatment resources (including options for HIV testing) in the local area. Patients will be told they show signs of risk associated with alcohol use in that they scored above a cut-score for our alcohol screen, and that they reported recently engaging in sexually risky behaviors. The staff person will advise patients that reducing their alcohol use, and illicit drug use when relevant, and using condoms is advised. BA will take approximately 5 minutes.
  Other Names: BA
  Arms: Brief Advice

SUMMARY:
This brief alcohol and sexual risk taking intervention has the potential to influence the public health by reducing alcohol use and sexual risk taking behavior in individuals who are seeking treatment in an Emergency Department.

DETAILED DESCRIPTION:
Linkages between alcohol use and HIV/sexual risk behaviors have been observed in multiple groups and each behavior has been successfully treated individually. Indeed, some studies suggest these behaviors can be successfully treated together. The Emergency Department (ED) provides a venue through which many patients with multiple risks are treated. Yet, to date no study has addressed these behaviors together in an ED, where admission may represent an opportunistic moment when patients are particularly willing to discuss these risky behaviors. Motivational Interviewing (MI) has demonstrated promise with alcohol risk in the ED in several of our previous studies, and has shown promise with sexual risk populations as well. Accordingly, this study (N=302) will address whether a one session multiple risk MI can more effectively decrease and maintain reduction in alcohol use, alcohol related problems, and sexual risk taking following discharge from the ED than Brief Advice (BA). Baseline, MI Session 1 and BA will be administered in the ED. Follow-ups will be conducted at 3, 6 and 9 months. This project will allow us to address the next phase of our program of research that has been designed to develop easily disseminable treatments for high-risk populations in medical settings. This study will also address potential mediators (motivation to change risk taking, self-efficacy) of MI effects. We will also examine whether reductions in sexual risk associated with MI compared to BA are accounted for by reduced drinking. A tertiary aim will examine the moderating effect of co-occurring substance use on outcomes. The cost-effectiveness of the interventions will also be addressed. Thus, this study will address two significant Public Health problems and provide significant information about MI mechanisms that may be relevant to the treatment community.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients older than 18 who receive medical care in the ED *score positive (> 8 for males; > 6 for females) for harmful alcohol use on the AUDIT screening questionnaire and report past 3-month binge drinking

  * be sexually active (past 6 months)
  * endorse any past-year sex-risk behavior criterion, including:

    * having more than one sexual partner
    * having sexual intercourse without a condom
    * consuming alcohol prior to or during sex
    * sing illicit drugs (or using licit drugs to get high) prior to or during sex.

Exclusion Criteria:

* Patients under the age of 18; Patients in a mutually monogamous relationship for longer than 1 year will be excluded unless either the patient or his/her partner are HIV+ or has unknown HIV status. Other exclusion criteria include:

  * scoring below 18 on a mini-mental status exam
  * no verifiable address
  * plans to move outside a 45-mile radius within the follow-up period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2011-05; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Monti, PhD, Principal Investigator — Brown University; Nadine R Mastroleo, PhD, Study Director — Brown University
Locations (3):
- United States (3):
  - Memorial Hospital of Rhode Island, Pawtucket, Rhode Island
  - Brown University Center for Alcohol and Addiction Studies, Providence, Rhode Island
  - Kent Hospital, Warwick, Rhode Island

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Conducted in two hospital Emergency Rooms in Rhode Island. Conducted between May 2011 and November 2013
Pre-assignment Details: 400 patients consented, 23 were lost prior to randomization, 5 withdrew from study prior to randomization, 45 did not completed the interventions
Period: Overall Study
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Started | 184 | 188
Completed | 154 | 173
Not Completed | 30 | 15
Not completed — Withdrawal by Subject | 7 | 0
Not completed — did not complete intervention | 23 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice | Total
Number analyzed (Participants) | 184 | 188 | 372
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 184 | 188 | 372
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.4 (9.1) | 30.0 (9.4) | 29.19 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 95 | 199
  Male | 80 | 93 | 173
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 184 | 188 | 372
Time-line Follow-back Alcohol and Sex (30 day) [Mean (Standard Deviation); unit: Days] — Tool used to retrospectively assess drinking and sexual behavior over the previous 30 days.
  Days | 5.8 (7.3) | 5.9 (6.8) | 5.9 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Alcoholic Drinks Consumed Per Week
Description: Number of standard alcoholic drinks consumed in the past month
Time Frame: 3 month
Population: 13 and 12 participants did not complete the assessment in the BMI and BA groups respectively
Measure: Mean (Standard Deviation); unit: Drinks per week
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Number analyzed (Participants) | 141 | 161
Drinks per week | 9.1 (11.5) | 16.5 (28.1)

2. Primary Outcome: Number of Alcoholic Drinks Consumed Past Month
Description: Number of standard alcoholic drinks consumed in the past month
Time Frame: 6-months
Population: 7 participants in each group did not complete the assessment.
Measure: Mean (Standard Deviation); unit: Drinks per month
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Number analyzed (Participants) | 147 | 166
Drinks per month | 9.2 (12.4) | 12.6 (17.9)

3. Primary Outcome: Number of Alcoholic Drinks Consumed Past Month
Description: Number of standard alcoholic drinks consumed in the past month
Time Frame: 9-months
Population: 5 and 9 participants did not complete the assessment in the BMI and BA groups respectively
Measure: Mean (Standard Deviation); unit: Drinks per month
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Number analyzed (Participants) | 149 | 164
Drinks per month | 8.4 (11.6) | 12.1 (17.6)

4. Primary Outcome: Number of Days Engaged in Risky Sex in the Past Month
Description: Number of days engaged in risky sex during the past month (condomless sex)
Time Frame: 3-months
Population: 13 and 12 participants did not complete the assessment in the BMI and BA groups respectively
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Number analyzed (Participants) | 141 | 161
Days | 0.8 (2.6) | 1.3 (4.0)

5. Primary Outcome: Number of Days Engaged in Condomless Sex in the Past Month
Description: Number of days engaged in compless sex during the past month
Time Frame: 6-months
Population: 7 participants in each group did not complete the assessment.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Number analyzed (Participants) | 147 | 166
Days | 0.7 (2.6) | 1.7 (4.9)

6. Primary Outcome: Number of Days Engaged in Condomless Sex in the Past Month
Description: Number of days engaged in condomless sex during the past month
Time Frame: 9-months
Population: 5 and 9 participants did not complete the assessment in the BMI and BA groups respectively
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Number analyzed (Participants) | 149 | 164
Days | 0.7 (2.9) | 0.9 (3.3)

ADVERSE EVENTS:
Arm/Group | Brief Motivational Intervention (BMI) | Brief Advice
Serious Adverse Events (participants affected / at risk) | 0/184 | 0/188
Other Adverse Events (participants affected / at risk) | 0/184 | 0/188

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No